CLINICAL TRIAL: NCT03944031
Title: Assessment of Brain O-GlcNAcase (OGA) Enzyme Occupancy After Single Oral Doses of LY3372689 as Measured by Positron Emission Tomography (PET) With the Radioligand [18F]LSN3316612 in Healthy Subjects
Brief Title: A Study of the Effects of LY3372689 on the Brain in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17220; I9X-MC-MTAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-02; First posted 2019-05-09 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04-15

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LY3372689 + [18F]LSN3316612 (Experimental): LY3372689 administered orally followed by [18F]LSN3316612 PET tracer administered intravenously (IV) approximately 2 - 72 hours later.
  Interventions: Drug: LY3372689; Diagnostic Test: [18F]LSN3316612

INTERVENTIONS:
Drug: LY3372689 — Administered orally.
Diagnostic Test: [18F]LSN3316612 — Administered IV.
  Other Names: [18F]MNI-1068

SUMMARY:
This study uses imaging to evaluate how LY3372689 binds to a protein in the brain. This study will be conducted in healthy participants and will last up to approximately 25 days after enrollment. Screening must be completed within 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females who cannot get pregnant
* Have a body mass index (BMI) of at least 18.5 kilogram per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study
* Have veins and arteries suitable for protocol required blood sampling

Exclusion Criteria:

* Have a history of head injury or contraindications to undergoing magnetic resonance imaging (MRI) examination
* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Smoke more than the equivalent of 10 cigarettes per day and are unwilling to stop smoking for study procedure
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate or could interfere with understanding the results of the study
* Have long exposure to sunlight routinely or use tanning beds regularly
* Participate in regular vigorous exercise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Percent O-GlcNAcase (OGA) Enzyme Occupancy (EO) | Predose Scan (Days -14 to -1)
  Percent OGA EO
Percent OGA EO | Postdose Scan 1 (Days 1 - 4)
  Percent OGA EO
Percent OGA EO | Postdose Scan 2 (Days 2 - 4)
  Percent OGA EO

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Invicro, Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No